CLINICAL TRIAL: NCT04284007
Title: Intravenous Versus Perineural Dexamethasone in Interscalene Nerve Block With Levobupivacaine for Shoulder and Upper Arm Surgeries
Brief Title: Intravenous Versus Perineural Effect Dexamethasone in Interscalene Nerve Block With Levobupivacaine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MFM_IRB, MS.18.03.65 -
Record Dates: First submitted 2019-12-28; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perineural levobupivacaine with intravenous saline (Active Comparator): Patients will receive levobupivacaine plus saline in interscalene brachial plexus block in addition to intravenous saline.
  Interventions: Drug: Perineural levobupivacaine
- Perineural dexamethasone in addition to levobupivacaine (Experimental): Patients will receive levobupivacaine-dexamethasone in interscalene brachial plexus block plus intravenous saline.
  Interventions: Drug: Perineural dexamethasone in addition to levobupivacaine
- Intravenous dexamethasone with perineural levobupivacaine (Experimental): Patients will receive levobupivacaine plus saline in interscalene brachial plexus block in addition to intravenous dexamethasone.
  Interventions: Drug: Intravenous dexamethasone with perineural levobupivacaine

INTERVENTIONS:
Drug: Perineural levobupivacaine — Patients will receive 20 ml of 0.25% levobupivacaine plus 2ml saline in interscalene brachial plexus block plus 10 ml intravenous saline.
  Arms: Perineural levobupivacaine with intravenous saline
Drug: Perineural dexamethasone in addition to levobupivacaine — Patients will receive 20 ml of 0.25% levobupivacaine plus 4mg dexamethasone diluted in 2 ml saline in interscalene brachial plexus block plus 10 ml intravenous saline.
  Arms: Perineural dexamethasone in addition to levobupivacaine
Drug: Intravenous dexamethasone with perineural levobupivacaine — Patients will receive 20 ml of 0.25% levobupivacaine plus 2ml saline in interscalene brachial plexus block plus 4 mg intravenous dexamethasone diluted in 10 ml saline.
  Arms: Intravenous dexamethasone with perineural levobupivacaine

SUMMARY:
Interscalene brachial plexus block can be used as an additive to general anaesthesia or as the primary anaesthetic for shoulder surgeries for pain management.

The investigators compared the effect of perineural versus intravenous dexamethasone on the prolongation of the action of levobupivacaine in ultrasound guided interscalene block for shoulder and upper arm surgeries.

DETAILED DESCRIPTION:
Dexamethasone had been shown to prolong the duration of postoperative analgesia when given as an adjuvant for peripheral nerve blocks.

The investigators compared the effect of perineural versus intravenous dexamethasone on the prolongation of the action of levobupivacaine in ultrasound guided interscalene block for shoulder and upper arm surgeries.

The study hypothesized that adding perineural dexamethasone to levobupivacaine in ultrasound guided interscalene block may be more superior to adding intravenous dexamethasone to levobupivacaine and levobupivacaine alone in shoulder and upper arm surgeries as regard analgesic effect, duration of analgesia and hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status grade I and grade II.

Exclusion Criteria:

* Patient refusal.
* Neuromuscular diseases (as myopathies, myasthenia gravies, …...)
* Hematological diseases, bleeding or coagulation abnormality.
* Psychiatric diseases.
* Local skin infection
* Sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2
* contralateral phrenic palsy
* pneumothorax
* pneumectomy
* severe COPD

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | for 24 hour postoperatively
  as measured by time to first analgesic requirement.

SECONDARY OUTCOMES:
Onset of Sensory block | For 30 min after injecting local anesthetic
  Patients will be closely observed until 30 minutes after the end of local anesthetic injection. Block success will be defined as loss of sensation to pinprick in the C4 and C5 sensory dermatome distribution measured 30 minutes after the end of local anesthetic injection. sensory block will be assessed by pin prick test using a 3point scale: • Grade 0 = Normal sensation.
  * Grade 1 = loss of sensation to pin prick (analgesia).
  * Grade 2 = loss of sensation to touch (anaesthesia). Onset time for sensory block will be defined as the time interval between the end of local anaesthesia administration and complete sensory block (score 2).
Duration of sensory block | within 24 hours after the surgery.
  defined as the time interval between complete sensory block (score 2) and complete resolution of anaesthesia on all nerves (score 0)
Onset time of motor block | For 30 min after injecting local anesthic
  Motor block will be determined according to the modified Bromage scale:
  * Grade 0 = Normal motor function with full flexion and extention of elbow.
  * Grade 1 = Decrease motor power.
  * Grade 2 = Complete motor block. Onset time of motor block will be defined as the time interval between end of local anaesthetic administration and complete motor block (grade 2).
Duration of motor block | within 24 hours after the surge
  defined as the time interval between complete motor block (score 2) and complete recovery of motor function of the arm (score 0).
Intraoperative Heart rate changes | For 3 hours after surgery
  Heart rate changes
Intraoperative Mean arterial blood pressure changes | For 3 hours after surgery
  Mean arterial blood pressure changes
Intraoperative analgesic consumption | For 3 hours after surgery
  the intraoperative analgesic dose consumption would be calculated The investigators can use fentanyl as analgesic if the patient required during the surgery ( 50-100 mic)
Postoperative heart rate changes | For one hour after admission to the postoperative anesthesia care unit
Postoperative Mean arterial blood pressure changes | For one hour after admission to the postoperative anesthesia care unit
Postoperative peripheral oxygen saturation changes | For one hour after admission to the postoperative anesthesia care unit
Pain score | Pain after surgery will be assessed using VAS at 1,2,6,12 and 24 hours.
  The VAS is represented with straight line with one end has the anchor " no pain" and it takes 0, while the other end of the line has the anchor " pain as bad as it could be" and it takes 10.
  The patient will receive the rescue analgesic when the score is more than 4)
Total analgesic need and the onset of first intravenous analgesia | After transportation of the patient from PACU up to 24 hours postoperative.
  Total analgesic need to rescue analgesic (pethidine) calculated by mg. And the onset of time for first intravenous analgesia during the 24 hours postoperative by hours.
Patient satisfaction: 2-point scale | first 24 hours postoperatively
  concerning the procedure is assessed using a 2-point scale (1= satisfied, I would want the same anesthesia / analgesia method for the next surgery, 2= unsatisfied, I would want a different anesthesia / analgesia method for the next surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Nahla S El-Ebahnsawy, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Hazem E Moawed, MD, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The raw data
Supporting Information: CSR
Time Frame: from January 2020 to December 2020
Access Criteria: Raw data and results with the registry